CLINICAL TRIAL: NCT02983357
Title: Long Term Outcome Follow-up of Glenoid Anchor Peg Component Fixation Utilizing Autologous Bone Graft in Total Shoulder Arthroplasty.
Brief Title: Long Term Outcomes Follow-up of Glenoid Anchor Peg Component Fixation
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0435-16-FB
Record Dates: First submitted 2016-11-04; First posted 2016-12-06 (Estimated); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Arthritis
Keywords: Shoulder Arthroplasty; glenohumeral arthritis
MeSH Terms: conditions — Arthritis | interventions — X-Rays; Restraint, Physical; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case Series Study: Subjects who received a total shoulder replacement with an anchor peg glenoid and autologous bone grafting at the department of Orthopaedic Surgery at University of Nebraska Medical Center / Nebraska Medicine and are now at least 9 years out from surgery.
  Interventions: Radiation: CT, X-Ray; Other: Physical assessment; Other: Questionnaire

INTERVENTIONS:
Radiation: CT, X-Ray — 2 anterior-posterior (AP) radiographs of the glenohumeral joint, one in internal rotation and the other in external rotation, along with axillary lateral films, will be completed of the affected operated shoulder. Also, a computed tomographic scan without contrast performed of same shoulder.
Other: Physical assessment — Physically evaluate for shoulder function and pain using American Shoulder Elbow Score (ASES) Constant score and the Simple Shoulder Test to obtain specific shoulder functional, motion,and strength outcomes.
Other: Questionnaire — Rand Short Form Health Survey (Rand SF-36) which is a patient completed quality of life measurement

SUMMARY:
The purpose of this study is to investigate if the use of autologous bone graft around the anchor-peg glenoid prosthesis correlates with (1.) bony apposition on computed tomography scans, (2.) decreased radiolucent lines, (3.) a decrease in component loosening, and (4.) better functional outcomes. Investigators hypothesize that a glenoid anchor peg component fixation utilizing autologous bone graft in Total Shoulder Arthroplasty (TSA) will have a lower incidence of glenoid loosening and that the absence of radiolucent lines will correlate with excellent shoulder function. Glenoid component loosening remains a major concern following total shoulder arthroplasty and is the man reason for failure. Despite positive findings in the investigators previous study (same population at a minimum of 2 year post operative follow up), it is reasonable that loosening rates could increase with longer follow-up. This study will be a minimum of 7 year post operative follow up.

DETAILED DESCRIPTION:
Long term outcome follow-up of glenoid anchor peg component fixation utilizing autologous bone graft in total shoulder arthroplasty. This research will be a case series study to evaluate the adequacy of fixation and functional outcome of the glenoid anchor peg following autologous bone grafting around the prosthesis at the time of implant. Eligibility criteria are subjects,who were treated at the Department of Orthopaedic Surgery at University of Nebraska Medical Center and Nebraska Medicine, with a total shoulder replacement using an anchor peg glenoid and autologous bone grafting, and who are now at least 9 years out from surgery. Each subject will be evaluated and this will include having three plain radiographs of the operated shoulder of which 2 will be true anterior-posterior (AP) radiographs of the glenohumeral joint, one in internal rotation and the other in external rotation, along with axillary lateral films. In addition, the subject will have a computed tomographic (CT) scan, without contrast dye, to examine the shoulder. One of the study personnel will use the Constant Score and Simple Shoulder Test to obtain specific shoulder functional, motion, and strength outcomes as well as pain assessment. A patient completed questionnaire, Rand Short Form Health Survey, (Rand SF-36) will be obtained to look at association with general health status. Investigators hypothesize that there will be a low incidence of glenoid loosening with a TSA (total shoulder arthroplasty) using an anchor peg glenoid and autologous bone grafting. In addition, investigators suggest that the absence of radiolucent lines will correlate with excellent shoulder function. A study was previously completed at our facility on same population at a minimum of 2 year follow up. At that time, and despite more than 10 years of widespread clinical use, no radiographic or clinical data existed regarding this unique component type. The findings from this prior study indicated that total shoulder arthroplasty (TSA) utilizing minimal glenoid peripheral peg cement and autologous reamings placed between radial fins of the central peg allowed host bone incorporation for the central peg and that better bone incorporation imparted fewer overall peg lucencies. The study findings were accepted for presentation at The American Academy of Orthopaedic Surgeons, 2010, New Orleans. Despite these positive findings, loosening rates could increase farther out from surgery, hence the purpose for the current proposed longer follow up study which is evaluation at a minimum of 9 years post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who received a total shoulder replacement with an anchor peg glenoid and autologous bone grafting at the department of Orthopaedic Surgery at University of Nebraska Medical Center / Nebraska Medicine and are now at least 9 years out from surgery.

Exclusion Criteria:

* Subjects who are unable to comprehend the consent form information. Pregnant women will be excluded from the study.

Ages: 44 Years to 94 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This research is a case series study to evaluate the adequacy of fixation and functional outcome of the glenoid anchor peg following autologous bone grafting around the prosthesis at the time of implant.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with bone presence between radial fins of the glenoid component's central peg measured by thin CT scans and using Yian CT-based radiolucency scores. | Day One
  CT

SECONDARY OUTCOMES:
Number of patients with glenoid component radiolucencies as measured by plain radiographs using Lazarus radiolucency scores for each. | Day One
  plain radiograph

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Teusink, MD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No